CLINICAL TRIAL: NCT03268564
Title: An Evidence-based Knowledge Transfer Program Promoting HIV Self-testing With Real-time Online Counseling for Men Who Have Sex With Men in Hong Kong
Brief Title: Promoting HIV Self-testing With Real-time Online Counseling for MSM in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KPF16ICF10
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Uptake of HIVST-online

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIVST-online promotion (Experimental): Health promotion for those who are not users of previous HIVST-online services (i.e. not "re-testers"):
  1. Viewing a promotion video and a demonstration video
  2. Brief motivational interviewing through telephone
  3. Visiting the HIVST-online webpage
  4. Receiving a free self-testing kit and follow-up reminders
  Health promotion for re-testers:
  1. Viewing a promotion video and a demonstration video
  2. Visiting the HIVST-online webpage
  3. Receiving a free self-testing kit and follow-up reminders
  Interventions: Behavioral: HIVST-online promotion

INTERVENTIONS:
Behavioral: HIVST-online promotion — Health promotion for those who are not users of previous HIVST-online services (i.e. not "re-testers"):
  1. Viewing a promotion video and a demonstration video
  2. Brief motivational interviewing through telephone
  3. Visiting the HIVST-online webpage
  4. Receiving a free self-testing kit and follow-up reminders
  Health promotion for re-testers:
  1. Viewing a promotion video and a demonstration video
  2. Visiting the HIVST-online webpage
  3. Receiving a free self-testing kit and follow-up reminders

SUMMARY:
Objectives To evaluate the efficacy of a program promoting HIV self-testing (HIVST) with online real-time counselling (HIVST-online) among men who have with men (MSM) in Hong Kong.

Participants Inclusion criteria are: i) Hong Kong Chinese speaking males aged ≥ 18 years old, ii) self-report having had anal sex with at least one man in the last six months, iii) willing to leave contacts (mobile phone and/or social media account), and iv) having access to online face-to-face communication tools like Line, Skype, or Facetime. Those having been diagnosed as HIV positive will be excluded.

Design A total of 350 eligible MSM will be recruited and invited to participate the program, including 120 HIVST-online users in a HMRF project (ref#11120791) (re-testers), and 230 new prospective HIV testers (new-testers) through outreaching at gay venues (bars and saunas), internet and social media, and referrals made by participants.

A brief baseline telephone survey will be conducted among all participants they are exposed to the components of the health promotion program. All participants will be followed up at Month 6 by phone/social media for outcome and process evaluation.

Main outcome measures The primary outcome is whether the participant has taken up our HIVST-online service during a 6-month follow-up period. This behavioural outcome will recorded objectively by the HIVST administrators. Among those who had not taken up HIVST at Month 6, they will be contacted by social media to ask a few questions to assess secondary outcomes, which include: 1) whether having taken up any form of HIV testing other than HIVST-online and 2) intention to take up HIVST-online or other forms of HIV testing in the next six months. Process evaluation of the health promotion components (e.g., online video, MI, and project webpage) and the HIVST-online service (e.g., delivery of the HIVST kits, appointment making with HIVST administrators, pre- and post-test counseling) will also be conducted.

DETAILED DESCRIPTION:
Objectives The investigators had developed an innovative home-based HIVST service (HIVST-online), which includes mailing a free HIVST kit and providing online real-time instructions and pre-test/post-test counseling via online live-chat applications to users

The objectives of this study are:

1. To promote men who have sex with men (MSM) who have never used the HIVST-online to use it for the first time.
2. To promote MSM who have used to HIVST-online to use it again.

Methods Target participants and recruitment

1. A total of 350 eligible MSM will be recruited and invited to take up the HIVST-online service. Inclusion criteria are: i) Hong Kong Chinese speaking males aged ≥ 18 years old, ii) self-report having had anal sex with at least one man in the last six months, iii) willing to leave contacts (mobile phone and/or social media account), and iv) having access to online face-to-face communication tools like Line, Skype, or Facetime. Those having been diagnosed as HIV positive will be excluded.
2. As a continuation, the 172 MSM who have used the HIVST-online service in our previous project will be invited to use HIVST-online again if they remain sexually active, as international recommendations suggest that sexually active MSM should take up HIV testing on a regular basis (e.g. once every six months). Modifications of the promotion messages will be made for these re-testers.
3. The target is to contact at least 70% of the 172 testers (n=120) and have 70% performing HIVST-online again (n=84). Therefore, the collaborating NGO will recruit about 230 new prospective HIV testers through outreaching at gay venues (bars and saunas), internet and social media, and referrals made by participants.

Health promotion Provision of health promotion of HIVST-online to prospective testers who are not users of previous HIVST-online services (i.e. not "re-testers")

Prospective testers, who are not "re-testers", will be sent via social media a link to access a webpage created for this project. They will then be exposed to the following components of health promotion which have shown to be effective in our previous project:

1. Viewing a promotion video and a demonstration video: Through the webpage, they will access an online video of about seven minutes in length promoting HIVST-online. The video had been used effectively in the previous HMRF HIVST-online project. The carefully design contents were guided by Health Belief Model. For instance, health communication messages are presented to increase viewers' perceived susceptibility of HIV infection and perceived benefit of HIVST-online. As the Social Cognitive Theory suggests that observational learning is effective in inducing health-related behaviors, the video also includes short testimonials about good experiences of HIVST-online made by a peer HIVST-online user. Another video demonstrating the use of HIVST (two minutes) will be sent to prospective participants; such a video is available from the ongoing project. Knowing that HIVST is easy to use would increase perceived confidence and hence self-efficacy (a Health Belief Model construct) in taking up HIVST-online.
2. Brief motivational interviewing (MI): The MI will be provided over phone or via social media by the research assistant(s) upon appointment and packaged as 'explaining the program' to the MSM interested in considering HIVST-online.
3. Visiting the HIVST-online webpage: The aforementioned videos can be accessed via this webpage. (i) Besides, it will contain a description of the project, knowledge and benefit of the HIVST, contact of the project team (phone, social media, and email), and information about HIV that promotes perceived susceptibility and perceived severity (constructs of the HBM). (ii) A discussion forum will be created to contain positive feedbacks of previous HIVST-online users (e.g. process evaluation of the previous RCT project), and those given by users of the proposed project. These testimonials provide cue to action (a construct of the Health Belief Model) and create a new subjective norm (a construct of the Theory of Planned Behavior) supporting the use of HIVST-online. As an incentive, a lucky draw will be made to those who leave encouraging comments to this forum. (iii) Participants and project team will add 'LIKE' or further comments to the webpage. (iv) Participants may post their questions in private, which will be answered by the project staff.
4. Receiving a free self-testing kit: Through phone and/or social media interactions, prospective users will provide a mailing address, and the investigators will send them a free HIVST kit (Aware TM Oral) in a plain envelope without any identification of the project. Participants will be given two alternative options for receiving the HIVST kit: 1) the investigators can warp the HIVST kit in a parcel without any identification of the project and send it to a Seven-Eleven store suggested by the participant by express. It is a common practice for people in HK to pick up their express from such stores. Upon receiving the express, a reminder SMS will be sent to the recipient by the store. Participants can pick up the parcel by showing the SMS they received without any additional charge; 2) the kit will be dispatched to them by volunteers. Receiving the test-kit is a strong cue to action (Health Belief Model, HBM) that may induce action. The practice was implemented smoothly in our HMRF project, for which we sent out about 200 self-test kits and most of those receiving the kit took up HIVST-online. The mailing of a free kit also removes logistic barriers required to buy or to collect a self-testing kit and cost concern (HBM). HIV rapid testing now being provided by the local NGOs and the government are also free of charge.
5. Follow-up reminders: Up to three weekly reminders will be sent by SMS/social media to those who had been sent a HIVST kit but have not registered for taking up HIVST-online (cue to action of the HBM). A hotline number answered by the research assistant will also be made available for those who need to discuss with us about their concerns.

Provision of health promotion of HIVST-online to "re-testers" As compared to the health promotion components for prospective testers who are not "re-testers", the "re-testers" will be exposed to a new and modified promotion video designed for them. Other components, such as the demonstration video, the project webpage, request for spreading the health promotion messages, receiving the free HIVST kits and follow-up reminders will be similar. As those who had used HIVST-online in the past have already shown motivation in using the service, they will not receive MI.

Actual implementation of the HIVST-online After being exposed to the various components of health promotion afore-mentioned, those MSM who decide to take up HIVST-online will contact the investigators and initiate the testing service. The following steps, which have been taken in the previous HMRF project, will be processed.

1. Testers will make an appointment with the investigators by phone/social media after they have received the HIVST kits by mail.
2. Through a communication tool (e.g., Line, Skype, Facetime or Whatsapp), the HIVST administrator will explain to the participants in detail how to use the HIVST. If necessary, the aforementioned demonstration video will be sent again to the testers. It is guaranteed that all information will be kept confidential. Participants are anonymous and do not need to show their faces if desired and no taping will be made.
3. The standard-of-care pre-test (risk assessment) and post-test counseling (e.g., interpretation of testing results and HIV prevention) of the HTC service will be implemented by a HIVST administrator (NGO staff), who will be trained by the HIVST administrator of our previous HMRF project.
4. The administrator will guide the tester to use the oral fluid based HIVST kit correctly. The HIVST kit to be used in this study (AwareTM Oral) is a brand of the Calypte Biomedical Corporation of the U.S., and is being manufactured by a subsidiary company of the Calypte Biomedical Corporation in Beijing. It has a proven sensitivity/specificity of >99.8% and has been approved for marketing by the State of Food and Drug Administration (SFDA) in China. It is now being used by CDC in China nationwide. This kit is available online at a price of 200HKD. The project team can obtain the kits at a discounted price at 80HKD per kit (liaison has been made with the manufacturer).
5. It takes about 20 minutes to know about the screening result. The entire testing and counseling process will take about 60 minutes, which is comparable to that needed for a traditional HTC in NGO or governmental clinic.
6. Those screened positive will be given immediate online psychological support. It will be emphasized that they have to take up a free confirmatory HIV antibody testing to be offered by the Department of Health. Referrals will be made whenever needed. The investigators may accompany them to visit the NGO (AIDS Concern) or the Department of Health if desired.

Evaluation Baseline survey A brief anonymous telephone survey will be conducted among all participants before they are exposed to the health promotion components of the program.

1. Background variables: 1) socio-demographic characteristics, 2) sexual orientation, 3) sexual behaviours in the last three months (type of male sex partners and female sex partners, and frequency of unprotected anal sex) and 4) substance use before/during sexual intercourse in the last three months.
2. HIV testing history: 1) HIV testing in lifetime and in the last three years, 2) types of HIV testing utilized in the last three years and in the last six months, and 3) behavioral intention to use any and specific types of HIV testing in the next six months. For re-testers, they will be asked additional questions about their satisfactory of the HIVST-online service provided by previous HMRF project.
3. Perceived risk of HIV infection in the next six months
4. Perceptions related to HIV self-testing: 1) positive attitudes toward HIV self-testing (e.g., convenient, privacy, etc.), 2) negative attitudes toward HIV self-testing (e.g., difficulty to interpret testing results by oneself, inadequate accuracy, etc.), 3) perceived subjective norm related to HIV self-testing (e.g., whether significant others would support them using HIV self-testing), 4) perceived behavioral control in using HIV self-testing, 5) behavioral intention to use HIV self-testing under different scenarios, 6) perceived importance of online real-time counseling supporting HIV self-testing and 7) preference of HIV self-testing kits (blood based or oral fluid based).

Month 6 follow-up evaluation Participants will be followed up by phone or social media for outcome and process evaluation.

The primary outcome is whether the participant has taken up our HIVST-online service during a 6-month follow-up period. This behavioral outcome is recorded by us objectively. Among those who had not taken up HIVST at Month 6, they will be contacted by phone/social media to ask several brief questions to assess secondary outcomes, which include: 1) whether having taken up any form of HIV testing other than HIVST-online and 2) intention to take up HIVST-online or other forms of HIV testing in the next six months.

Process evaluation All participants will be asked some questions through phone/social media as a process evaluation of the health promotion components (e.g., online video, MI, and project webpage). All testers of the HIVST-online will be asked additional questions rating their satisfaction of various aspects of the HIVST-online service (e.g., delivery of the HIVST kits, appointment making with HIVST administrators, pre- and post-test counseling).

ELIGIBILITY:
Inclusion Criteria:

* 1) Hong Kong Chinese speaking males aged ≥ 18 years old, 2) self-report having had anal sex with at least one man in the last six months, 3) willing to leave contacts (mobile phone and/or social media account), and 4) having access to online face-to-face communication tools like Line, Skype, or Facetime

Exclusion Criteria:

* Diagnosed as HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Taken up our HIVST-online service | 6 months
  Taken up our HIVST-online service during a 6-month follow-up period

SECONDARY OUTCOMES:
Taken up any form of HIV testing other than HIVST-online | 6 months
  Taken up any form of HIV testing other than HIVST-online during a 6-month follow-up period
Intention to take up HIVST-online or other forms of HIV testing | 6 months
  Intention to take up HIVST-online or other forms of HIV testing in the next six months

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong